CLINICAL TRIAL: NCT01967550
Title: A 4-week, Randomized, Double-blind, Multi-center, Vehicle-controlled, Parallel Group Study to Assess the Efficacy and Safety of Diclofenac Diethylamine 2.32% Gel for the Relief of Signs and Symptoms in Patients With Knee Osteoarthritis
Brief Title: Efficacy and Safety of Diclofenac DDEA 2.32 % in Patient Suffering From Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 194-P-308; 2012-004024-38 (EudraCT Number)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Symptomatic knee OA Kellgren-Lawrence grade 1-3
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — diclofenac diethylamine; di-N-desethylamiodarone; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- diclofenac diethylamine, DDEA 2.32% gel (Experimental): diclofenac diethylamine, DDEA 2.32% gel
  Interventions: Drug: diclofenac diethylamine, DDEA 2.32% gel
- Placebo (Placebo Comparator): Vehicle control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: diclofenac diethylamine, DDEA 2.32% gel
  Arms: diclofenac diethylamine, DDEA 2.32% gel
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of diclofenac DDEA 2.32 % in patient suffering from knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female ≥ 50 years old; 2. Symptomatic OA of one or both knees, according to ACR criteria, diagnosed at least 6 months previously; 3. Pain in either knee originates in the knee (not referred pain from other sites, such as hip or back) and no other cause of pain than knee OA; 4. Have used oral NSAIDs or COXIBs for the knee OA pain (including aspirin if ≥ 500 mg and used in this indication), at least one dose per day, for not less than 10 days out of the 14 days preceding the screening visit and also within the 24 hours preceding the screening visit; 5. Be able to tolerate rescue medication with only 500 mg paracetamol (APAP) taken in doses of 1-2 tablets up to a maximum of 6 tablets (3 grams) per day for the duration of the study

Exclusion Criteria:

- 1. Partial or total replacement of either knee joint, past or planned/expected during study duration.

2. OA of the knee due to other underlying conditions, such as gout, chondrocalcinosis, hemochromatosis, joint infections, neuropathia, or severe traumatic joint damage (however, common risk factors, such as obesity and past meniscectomy or ligament rupture and repair, are allowed); 3. History of systemic inflammatory (autoimmune) disease (rheumatoid arthritis, systemic psoriasis, systemic lupus erythematosus, systemic sclerosis, etc.) or laboratory values indicative of such disease with subsequent diagnosis by a physician; 4. Fibromyalgia within the previous year; 5. Allergy or asthma to diclofenac, APAP, aspirin, other NSAIDs or any of the ingredients in the gel (i.e. isopropyl alcohol, propylene glycol, or butylhydroxytoluene), or any other contraindication for the study drug or the rescue medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Bad Hersfeld
  - Berlin
  - Hamburg
  - Munich
  - Stockach

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date 04 Oct 2013 end date 05 May 2014
Period: Overall Study
Arm/Group | Diclofenac Diethylamine, DDEA 2.32% Gel | Placebo
Started | 153 | 151
Completed | 148 | 149
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Non Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Diethylamine, DDEA 2.32% Gel | Placebo | Total
Number analyzed (Participants) | 153 | 151 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.8) | 65.1 (8.5) | 64.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 99 | 196
  Male | 56 | 52 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 131 | 127 | 258
  Unknown or Not Reported | 22 | 24 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 153 | 150 | 303
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 153 | 151 | 304

OUTCOME MEASURES:

1. Primary Outcome: Measure: Pain On Movement (POM)
Description: POM will be assessed by subject on a 100 mm Visual Analog Scale (VAS). The VAS ranges from 0 to 100 with higher score indicating higher levels of pain.
Time Frame: 2 weeks
Population: The modified ITT (mITT) population excludes subjects in the ITT population who were incorrectly instructed by the investigator to treat only one knee. The mITT population is primary for the analysis of efficacy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac Diethylamine, DDEA 2.32% Gel | Placebo
Number analyzed (Participants) | 141 | 141
units on a scale | 42.9 (23.8) | 42.1 (23.5)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Diclofenac Diethylamine, DDEA 2.32% Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/151
Other Adverse Events (participants affected / at risk) | 48/153 | 47/151
OTHER ADVERSE EVENTS (reported when occurring in more than 0.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Diethylamine, DDEA 2.32% Gel (N=153) | Placebo (N=151)
Headache (Nervous system disorders) | 18 (18) | 18 (18)
Nasopharyngitis (Infections and infestations) | 4 (4) | 10 (10)
Contusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respioratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dental operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Conjonctivitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0)
Application site warmth (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Spinal Pain (General disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator